CLINICAL TRIAL: NCT04570397
Title: C5 Complement Inhbition Using Ravulizumab for the Treatment of COVID-19 Induced Thrombotic Microangiopathy
Brief Title: Ravulizumab and COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Andrew Michael Siedlecki, asistant professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 092420
Record Dates: First submitted 2020-09-29; First posted 2020-09-30 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Covid19; Thrombotic Microangiopathies; Acute Kidney Injury
MeSH Terms: conditions — COVID-19; Thrombotic Microangiopathies; Acute Kidney Injury | interventions — ravulizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional arm (Experimental): ravulizumab
  Interventions: Drug: Ravulizumab
- Control arm (No Intervention): patients in this arm will recieve standard care

INTERVENTIONS:
Drug: Ravulizumab — Patients will receive weight-based dosing of ravulizumab on Days 1, 5, 10, and 15 along with the standard care.
  Arms: Interventional arm

SUMMARY:
Ultomiris (Ravulizumab), is a monoclonal antibody that specifically targets terminal complement products and is proposed for the treatment of COVID-19 induced microvasculature injury and endothelial damage leading to thrombotic microangiopathy (TMA) causing acute kidney injury (AKI). Ravulizumab is to be used for participants with a confirmed diagnosis of COVID-19 who clinically or diagnostically present with deteriorating renal function. Ravulizumab causes immediate and sustained inhibition of the terminal complement cascade. The use of ravulizumab could ameliorate COVID-19 induced kidney injury due to TMA, shorten hospital stay, and improve the overall survival.

DETAILED DESCRIPTION:
The novel coronavirus (COVID 19) is responsible for the current pandemic with the numbers of diagnoses and fatalities rising daily. It is reported that of those requiring medical intensive care almost 49% will expire prior hospital discharge. The initial peak of hospitalized patients in Boston, MA occurred on April 15, 2020 however new presentations continue to manifest at a local and national level.

The exact pathophysiology is still not clear. There are various theories that explain the pathophysiology which includes but is not limited to direct viral damage via the angiotensin-converting enzyme 2 receptor, systemic inflammatory response with cytokine storm, and aggravated hypoxia.

Recently, it has been observed that signs and symptoms of severe COVID 19 describe complement-mediated TMA rather than the sepsis induced coagulopathy. This strengthens the hypothesis that complement inhibition by C5a inhibitor, Ultomiris (ravulizumab) could ameliorate COVID 19 induced TMA, improve renal function, shorten the hospital stay and reduce the overall mortality.

In those affected with severe or fatal COVID-19, there is evidence of end-organ damage with acute kidney injury which has heightened the interest in studying the excessive cytokine release and its overall effect in the form of multi-organ failure.

Ultomiris (Ravulizumab) is a long acting second generation monoclonal antibody against a terminal complement product C5a and is FDA approved for the treatment of Paroxysmal Nocturnal Hemoglobinuria (PNH) and atypical hemolytic uremic syndrome.The benefit of Ultomiris has not been clinically evaluated in COVID 19 induced TMA.

Recently, ravulizumab has been utilized in the setting of a phase 3 clinical trial for the treatment of COVID 19 induced pneumonia, acute lung injury and acute respiratory distress. As it binds to C5 and impedes the cleavage of C5 by C5 convertase to generate C5a and membrane attack complex, ravulizumab could possibly improve the renal function in COVID 19 induced TMA and potentially improve overall survival, due to similar pathophysiology in the microvasculature of the kidney. More so, studies are being conducted to determine renal and cardiovascular sequelae of COVID-19 infection, which further enhances the interest to closely examine and evaluate those patients presenting 30-60 days after COVID-19 infection with signs of renal failure. There remains an unmet clinical need to investigate this approach with a randomized controlled trial to determine if complement cascade inhibition can improve the clinical outcome for COVID 19 induced acute kidney injury as measured by improvement of renal function and decline in the overall morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Males or Females 18 years of age or above and weighing 40kg or above at the time of providing informed consent.
2. A clinical diagnosis of thrombotic microangiopathy will then be applied to include the following criteria: i) D-dimer > 100% the upper limit of the reference range and ii) serum creatinine >25% of the normal range or iii) >25% increase from patient's baseline serum creatinine.
3. Diagnosis of SARS-CoV-2 infection within 90 days prior to enrollment

Exclusion Criteria:

1. Participant is not expected to survive more than 24 hours.
2. Participant has an unresolved Neisseria Meningitides infection.
3. Hypersensitivity to murine proteins or to one of the excipients of ravulizumab.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-12-18 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Assess the efficacy of ravulizumab to ameliorate SARS-CoV-2 (COVID-19)-induced acute kidney injury manifesting as thrombotic microangiopathy. | 30 days
  50% improvement in estimated glomerular filtration rate compared to conventional therapy within 30 days of treatment for COVID-19-induced acute kidney injury.

SECONDARY OUTCOMES:
Evaluation of pharmacokinetics of ravulizumab in participants with COVID-19 | 120 days
  Evaluation of pharmacokinetics of ravulizumab in participants with COVID-19 Changes in ravulizumab concentration in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States